CLINICAL TRIAL: NCT06243068
Title: Improving Shared Decision-Making and Access to Non-Dialytic Treatment for People With Kidney Disease (The ExPAND Trial)
Brief Title: Expanding and Promoting Alternative Care and kNowledge in Decision-making Trial
Acronym: ExPAND
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: West Virginia University Research Corporation (Unknown); University of Bristol (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCR235148; IHS-2022C2-27678 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-12-20; First posted 2024-02-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease
Keywords: CKD; Alternative Treatment Plan; KDE; Kidney Disease Education; Palliative Care; Shared-Decision Making; Active Medical Management without Dialysis; AMCWD; Kidney Supportive Care; ESRD
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: We will use a repeated cross-sectional stepped wedge design with randomization at the practice level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educate and Engage (Experimental): Patients accrued and making treatment decisions while the clinic treating them is implementing Approach 1.
  Interventions: Behavioral: Educate and Engage
- Educate and Engage Plus Kidney Supportive Care Program (Experimental): Patients accrued and making treatment decisions while the clinic treating them is implementing Approach 2.
  Interventions: Behavioral: Educate and Engage Plus Kidney Supportive Care Program

INTERVENTIONS:
Behavioral: Educate and Engage — Nephrology practices implement a bundle in which they will encourage their patients to a) participate in a kidney disease education program providing a balanced presentation of all options including ATPs, b) use evidence-based patient decision aids that include ATPs, and c) engage in shared decision-making with staff who have been trained in communication skills and best practices.
  Arms: Educate and Engage
Behavioral: Educate and Engage Plus Kidney Supportive Care Program — In addition to bundle described under "Educate and Engage," nephrology practices offer a systematic program integrating primary palliative care to support patients and their families who choose any ATP. The program closely follows patients and their families on ATP with care coordination, symptom management, advance care planning, and psychosocial support to supplement usual care from their nephrologist.
  Arms: Educate and Engage Plus Kidney Supportive Care Program

SUMMARY:
The goal of this clinical trial is to compare two health system-based approaches for offering kidney failure treatment options to older patients with kidney failure, specifically, to ensure patients are actively involved in a shared decision making (SDM) process covering a full range of treatment choices and have meaningful access to that full range of choices. These include standard in-center or home dialysis as well as alternative treatment plans (ATPs): active medical care without dialysis, time-limited trial of dialysis, palliative dialysis, and deciding not to decide.

Approach 1 - Educate and Engage:

Nephrology practices encourage their patients to a) participate in a kidney disease education program providing a balanced presentation of all options including ATPs, b) use evidence-based patient decision aids that include ATPs, and c) engage in SDM with staff trained in communication skills and best practices.

Approach 2 - Educate and Engage Plus Kidney Supportive Care Program:

Nephrology practices add a primary palliative care program to support patients who choose ATPs and their families. The program provides care coordination, symptom management, advance care planning, and psychosocial support to supplement usual care from their nephrologist.

To compare the two approaches, the investigators will conduct a repeated, cross-sectional stepped wedge cluster randomized trial involving 20-25 chronic kidney disease clinics at 8 practice organizations around the United States.

Aim 1: Compare the effectiveness of Approaches 1 and 2 in a) increasing proportion of patients choosing ATP and b) reducing patient-reported decisional conflict about treatment.

Aim 2: Compare the patient and family experience of ATP care between Approaches 1 and 2 in terms of quality of life, services used, and end of life (EOL) experience. Aim 2a will focus on experience while patients are receiving an ATP. Aim 2b will describe the EOL experience.

Aim 3: Evaluate implementation of each approach through a mixed-methods design based on the expanded RE-AIM framework.

For Aims 1 and 2, researchers will collect information by chart review and surveys with patients and caregivers. For Aim 3, clinic administrators, clinical providers, and staff will complete pre- and post-test surveys at the beginning and end of each training.

DETAILED DESCRIPTION:
Detailed Description

Background: Over 130,000 patients with kidney failure start dialysis annually. Older patients constitute the fastest growing segment. Those who are frail or have other serious medical conditions may not live any longer with dialysis than without it. US healthcare policy has created a powerful "dialysis default," where virtually all patients with kidney failure who do not receive a transplant are treated with a standard dialysis regimen in a dialysis center regardless of whether it will help them live any longer or better. About 20% of patients regret the decision to start dialysis, yet non-dialysis alternatives are rarely offered to them. Most patients report they were unaware they had a choice about kidney failure treatment. Many older patients with kidney disease value independence over staying alive longer. Not aware of their patients' values, most nephrologists do not offer alternatives to standard dialysis such as active medical care without dialysis (AMCWD), a time-limited trial of dialysis (TLT), palliative dialysis, or deciding not to decide (DND) until a later date.

Similarly, these options, which the investigators have collectively labeled alternative treatment plans (ATPs), are rarely included in kidney disease education (KDE) sessions for patients funded by Medicare. Other countries-notably Australia, Canada, and the United Kingdom-have found that about 15% of older patients with kidney failure prefer AMCWD. These countries have created programs within their healthcare systems that integrate primary palliative care into care for patients who choose an ATP. These programs report excellent outcomes in terms of patient quality of life, care according to patient's wishes, and patient survival on average for over a year. These programs have shown it is possible to avoid complications at the end of life such as patients who wanted AMCWD being started on dialysis because their symptoms were not well managed. These programs provide an extra layer of support and prepare patients and families for when the patient's kidney failure worsens.

Shared decision-making (SDM) is recognized as the preferred approach to implementing patient-centered care and assuring that patients receive treatment that matches their goals. For over a decade, SDM has been recommended by nephrology professional societies before initiating dialysis. Despite the recommendation and preference for SDM of people with advanced chronic kidney disease (CKD), it remains poorly implemented, and observers have noted a powerful dialysis default with few perceived alternatives. There is an urgent need for strategies to increase adoption and implementation of SDM in nephrology practices and elsewhere in healthcare systems where CKD patients receive care.

Objective: The goal of this clinical trial is to compare two health system-based approaches for offering kidney failure treatment options to older patients with kidney failure. Specifically, the goal is to ensure patients with kidney failure are actively involved in a SDM process covering a full range of treatment choices and have meaningful access to that full range of choices. These include standard in-center or home dialysis as well as alternative treatment plans: active medical management without dialysis (AMCWD), time-limited trial of dialysis (TLT), palliative dialysis, and deciding not to decide (DND).

Interventions - Approach 1: Educate and Engage In this approach, nephrology practices implement a bundle in which the participants will encourage their patients to a) participate in a kidney disease education program providing a balanced presentation of all options including ATPs, b) use evidence-based patient decision aids that include ATPs, and c) engage in shared decision-making with staff who have been trained in communication skills and best practices.

Interventions - Approach 2: Educate and Engage Plus Kidney Supportive Care Program In this approach, nephrology practices continue to implement the Educate and Engage bundle and additionally, offer a systematic program integrating primary palliative care to support patients and their families who choose any ATP. The program closely follows patients and their families on ATP with care coordination, symptom management, advance care planning, and psychosocial support to supplement usual care from their nephrologist.

Study Design: To compare the two approaches, the investigators will conduct a repeated, cross-sectional stepped wedge cluster randomized trial (SW-CRT) involving 20-25 chronic kidney disease clinics at 8 practice organizations around the United States. Participating clinical sites will be randomly placed into one of three sequences. Each sequence consists of four 10-month time periods during which patients are accrued and followed for study outcomes. All practices begin by implementing Approach 1 (Educate and Engage). Practices then add Approach 2 (Kidney Supportive Care Program) at the assigned period based on their sequence. To minimize contamination in the primary analysis, we will exclude patients recruited during the 4 months before each sequence moves to Approach 2. These patients will be included in a sensitivity analysis. In the 4th study period, accrual of new patients will stop during a 4-month follow-up period (to collect primary outcomes) at the end of the study. Patients will receive the intervention based on the approach (condition) in which the site is enrolled at the time of accrual. When a practice site begins implementation of Approach 2, referral to the kidney supportive care program for patients considering ATPs will become standard care at that site. All patients still alive who chose ATPs in prior periods will be offered the option of receiving care from the newly organized supportive care program.

In addition to the primary SW-CRT comparing the two intervention approaches, the investigators will do a pre-post comparison of primary outcomes, comparing clinic practices at baseline with each of the interventions.

Aim 1: Compare the effectiveness of two approaches: 1) improved kidney disease education (KDE) and SDM or 2) improved KDE and SDM plus the creation of a kidney supportive care program in a) increasing proportion of patients choosing ATP and b) reducing patient-reported decisional conflict.

Aim 2: Compare the patient and family experience of an ATP between Approach 1 and Approach 2 in terms of quality of life, services used, and end of life (EOL) experience through medical record review and interviews with a sample of patients, family members, and caregivers. Aim 2a will focus on experience while patients are receiving an ATP (several months to several years). Aim 2b will describe the EOL experience.

Aim 3: Evaluate implementation of each intervention (Approaches 1 and 2) through a mixed-methods design based on the expanded RE-AIM framework, which integrates the Implementation Outcomes Framework by positing that the implementation outcomes acceptability (whether interventions are agreeable and satisfactory), appropriateness (perceived fit, relevance, and compatibility), and feasibility (extent to which interventions can be used successfully) are predictors of successful adoption, implementation, and maintenance. The ExPAND research team will cooperate with a separate tandem evaluation conducted by an independent evaluation team based at NORC.

Study Activities and Data Collection for Aim 1

* Patients 65 years of age or older will be enrolled when their eGFR drops below 30.
* Patients are invited to take a series of three surveys that include the Decision Conflict Scale, Knowledge Assessment Scale, and patient experience of shared decision-making using SDM-Q-9, CollaboRATE, and other assessments. The baseline survey (DCS-1) is taken at the time of enrollment. Follow-up surveys are conducted at Month 4 and Month 9 after enrollment.
* The research coordinator (RC) conducts a chart audit to look for advance care planning documentation and current treatment preference 4 months after enrollment.

Study Activities and Data Collection for Aim 2 - Patients who choose an ATP

* The RC conducts a monthly chart audit for each patient who chooses an alternative treatment plan. The audit assesses the number of clinic visits, hospitalizations, changes in treatment plans, and unplanned dialysis starts.
* A small open cohort of ATP patients and their family members/care partners are invited to participate in a longitudinal series of interviews about their experience of care under an ATP, starting at the time of treatment decision and continuing every 4 months until the end of the study or death of the patient.
* For ATP patients who die, the RC conducts a chart review to assess EOL service utilization and advance care planning.
* A purposeful sample of family members/care partners of ATP patients are invited to participate in bereavement interviews 4 months after patient death.

Study Activities and Data Collection for Aim 3

• Clinic administrators, clinicians, and staff are invited to participate in pre-and post-test surveys at beginning and end of training.

ELIGIBILITY:
Study Population 1: Person with CKD, cared for at participating clinic

Inclusion Criteria:

* Age 65 years or older
* Most recent eGFR <30 at time of screening AND meets practice site criteria for KDE referral
* Treatment naïve (no dialysis or kidney transplant prior to enrollment)

Exclusion Criteria:

* The patient is a transplant candidate.
* The current decrease in eGFR is thought to be due to an acute event.
* Education and initiation of shared decision-making process are not yet indicated for the patient, (per practice protocol and/or provider's judgment).

Exclusion Criteria for primary analysis:

- Insufficient decision making capacity (Outcomes for this group will be described separately.)

Exclusion Criteria for surveys and interviews:

* Insufficient decision making capacity
* Non-English and non-Spanish speaking
* Treating nephrologist/APP opts patient out (for example, if contraindicated for patient's health)

Study Population 2: Family member or caregiver of patient in Study Population 1

Inclusion Criteria:

* Family member or caregiver of Population 1 patient who has chosen alternative treatment plan
* 18+ years old
* English or Spanish speaking
* Cognitively able to participate in surveys/interviews

Study Population 3: Administrator, clinical provider, or staff at participating chronic kidney disease clinic

Inclusion Criteria:

- Currently practicing or employed at participating clinic

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients choosing Alternative Treatment Plans (ATP) | Month 4 after enrollment.
  Numerator: number of patients choosing an alternative treatment plan. Denominator: enrolled patients with decision-making capacity.
Decisional Conflict Scale score | Month 4 after enrollment.
  Decisional Conflict Scale (O'Connor, 1995) score at month 4 survey, adjusted for baseline score. Score ranges from 0 (no decisional conflict) to 100 (extremely high decisional conflict).

SECONDARY OUTCOMES:
Rating of CKD Knowledge Among Older Adults (Know-CKD) score | Four months after enrollment.
  Rating of CKD Knowledge Among Older Adults (Know-CKD) 4 months after initiation of treatment decision-making process. Decision-Aid for Renal Therapy (DART) Knowledge Assessment (Ladin et al., 2023). The DART survey contains 10 items scored on a 3 point scale, with 0 points given for an answer of yes, 2 for an answer of unsure, and 4 for an answer of no. The total score is the sum of the 10 items, multiplied by 2.5. The minimum score possible is 0 (no decisional conflict) and the maximum score possible is 100 (extremely high decisional conflict) (Month three score, adjusted for baseline score)
Shared Decision Making Questionnaire (SDM-Q-9) score | Month 4 after enrollment.
  9-Item Shared Decision Making Questionnaire (SDM-Q-9) score (Scholl, 2010). Score ranges from 0 (least SDM) to 45 (most SDM).
CollaboRATE score | Month 4 after enrollment.
  CollaboRATE score (Elwyn et al., 2013). Scores range from 0 (least SDM) to 9 (most SDM).
Patient reported decision regret | Month 9 after enrollment.
  Modification of dialysis decision regret (Saeed et al., 2020) : Do you regret your treatment decision? 5-point Likert scale from 1 to 5, with 1 being "no regret at all" and 5 begin "a lot of regret".
Advance care planning (ACP) documentation | Month 4 after enrollment.
  Complete ACP measure (Three elements present in chart: a surrogate, a goals of care discussion, and either an accessible advance directive or medical order such as POLST or DNR.)
Proportion of Active Medical Care Without Dialysis (AMCWD) patients who change to dialysis at any time | From date of initial treatment decision to date of changed treatment decision, start of dialysis, patient death or end of study, whichever came first, assessed up to 40 months.
  Proportion of patients who initially choose AMCWD who subsequently switch to dialysis (standard in-center hemodialysis, home dialysis, time-limited trial, or palliative).
Proportion of ATP patients who have an unplanned transition into dialysis | From date of initial treatment decision to date of changed treatment decision, start of dialysis, patient death or end of study, whichever came first, assessed up to 40 months.
  Proportion of patients who initially choose an ATP who subsequently have an unplanned dialysis start: defined as starting dialysis urgently in the hospital during an unscheduled admission.
End of Life intensity scale | Final 30 days of life, (60 days and 90 days for sensitivity analysis). Assessed 3 months after patient death.
  Modified scale adapted from Wong et al, 2012, based on health services received during the last month of life (dialysis, emergency department, hospital, ICU), and death in hospital. Scores range from 0-6 with a higher score indicating more intensive end-of-life care.
AMCWD & DND patients who initiate dialysis in the last month of life | Final 30 days of life, (60 days and 90 days for sensitivity analysis). Assessed 3 months after patient death.
  Of AMCWD & DND patients die during the study, proportion who used dialysis in last 30 days of life.
For ATP patients, advance care planning (ACP) documentation at time of death. | Time of death. Collected 3 months after patient death.
  Complete ACP measure (Three elements present in chart: a surrogate, a goals of care discussion, and either an accessible advance directive or medical order such as POLST or DNR.)
Proportion of eligible clinicians who engage patients in Shared Decision Making (SDM) | Reported monthly by site manager in monthly progress reports, assessed from start to end of study, up to 40 months
  Proportion of eligible clinicians who engage patients in SDM. Demographic representativeness will be also be described.
Proportion of eligible clinicians who increase the proportion of patients choosing ATP | Reported monthly by site manager in monthly progress reports, assessed from start to end of study, up to 40 months
  Proportion of eligible clinicians who increase the proportion of patients choosing ATP. Demographic representativeness will be also be described.
Proportion of eligible practice sites that offer Kidney Disease Education (KDE) | Reported monthly by site manager in monthly progress reports, assessed from start to end of study, up to 40 months
  Proportion of eligible practice sites that offer KDE. Demographic representativeness will be also be described.
Proportion of eligible practice sites that offer Kidney Supportive Care (KSC) program | Reported monthly by site manager in monthly progress reports, assessed from start to end of study, up to 40 months
  Proportion of eligible practice sites that offer KSC. Demographic representativeness will be also be described.

OTHER OUTCOMES:
McGill Quality of Life Part A Score | Starts after consent to participate in longitudinal interviews. Repeats every 4 months until first of project completion or patient death, assessed up to 40 months.
  McGill Quality of Life score (Cohen et al., 1997). Based on responses to Part A, scores range from 0 (very bad) to 10 (excellent). Repeated measure, reported by a convenience sample of patients and care partners who choose an ATP and participate in a longitudinal series of interviews.
ATP patient reports of experience of ATP care (qualitative) | Starts after consent to participate in longitudinal interviews. Repeats every 4 months until first of project completion or patient death, assessed up to 40 months.]
  Responses to open-ended questions about the experience of receiving care under an alternative treatment plan. Reported by a convenience sample of patients who choose an ATP and participate in a longitudinal series of interviews.
Caregiver reports of caregiving experience (qualitative) | Starts after consent to participate in longitudinal interviews. Repeats every 4 months until first of project completion or patient death, assessed up to 40 months.
  Responses to open-ended questions of experience caring for patients who have selected ATP. Reported by a convenience sample of caregivers who have consented to participate in a longitudinal series of interviews.
Hospice use by ATP patients | End of life. Collected by chart review 3 months after death.
  Among ATP patients, proportion of deaths with hospice care, length of use of hospice.
Proportion of eligible patients who enroll in the Kidney Supportive Care Program | Reported monthly by site manager in monthly progress reports, assessed from start to end of study, up to 40 months
  Proportion of eligible patients (patients who choose an ATP under Approach 2) who enroll in the Kidney Supportive Care Program. Demographic representativeness will be also be described.
Caregiver reports of their experience of end-of-life care (qualitative) | End of life. Bereavement interview conducted 4 months after patient death.
  Responses to open-ended questions of experience caring for patients who have selected ATP and have died. Reported by a convenience sample of caregivers who have consented to participate in a longitudinal series of interviews.
Decisional conflict scale subscale scores | Month 4 after enrollment.
  Decisional Conflict Survey subscale (O'Connor, 1995) scores at month 4 survey, adjusted for baseline score. Score ranges from 0 (no decisional conflict) to 100 (extremely high decisional conflict).

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - UCSF/Zuckerberg San Francisco General Hospital and Trauma Center-Nephrology, San Francisco, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Southeast Kidney Associates, Canton, Georgia
  - Southeast Kidney Associates, East Point, Georgia
  - St. Clair Nephrology, Shelby, Michigan
  - The Rogosin Institute Manhattan Eat Dialysis, New York, New York
  - Clinical Renal Associates, Exton, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Renal Disease Research Institute, Dallas, Texas
  - Renal Disease Research Institute, Fort Worth, Texas
  - Renal Disease Research Institute, Garland, Texas
  - Renal Disease Research Institute, Irving, Texas
  - North Texas Kidney Disease Associates, Lewisville, Texas
  - Renal Disease Research Institute, McKinney, Texas
  - Renal Disease Research Institute, Mesquite, Texas
  - North Texas Kidney Disease Associates, North Richland Hills, Texas
  - North Texas Kidney Disease Associates, Plano, Texas
  - Renal Disease Research Institute, Plano, Texas
  - Virginia Nephrology Group, Alexandria, Virginia
  - Virginia Nephrology Group, Arlington, Virginia
  - Virginia Nephrology Group, Fairfax, Virginia
  - West Virginia University Medicine, Fairmont, West Virginia
  - West Virginia University Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, the completely deidentified research data from this project will be deposited with the digital repository, the Patient-Centered Outcomes Data Repository (PCODR), of the Inter-university Consortium for Political and Social Research (ICPSR), University of Michigan to ensure that the research community has long-term access to the data. This is required by PCORI and included in consent forms.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Per PCORI guidelines
Access Criteria: Per PCORI guidelines

REFERENCES:
- [Background] Cohen SR, Mount BM, Bruera E, Provost M, Rowe J, Tong K. Validity of the McGill Quality of Life Questionnaire in the palliative care setting: a multi-centre Canadian study demonstrating the importance of the existential domain. Palliat Med. 1997 Jan;11(1):3-20. doi: 10.1177/026921639701100102. PMID 9068681
- [Background] Engelberg R, Downey L, Curtis JR. Psychometric characteristics of a quality of communication questionnaire assessing communication about end-of-life care. J Palliat Med. 2006 Oct;9(5):1086-98. doi: 10.1089/jpm.2006.9.1086. PMID 17040146
- [Background] Ladin K, Tighiouart H, Bronzi O, Koch-Weser S, Wong JB, Levine S, Agarwal A, Ren L, Degnan J, Sewall LN, Kuramitsu B, Fox P, Gordon EJ, Isakova T, Rifkin D, Rossi A, Weiner DE. Effectiveness of an Intervention to Improve Decision Making for Older Patients With Advanced Chronic Kidney Disease : A Randomized Controlled Trial. Ann Intern Med. 2023 Jan;176(1):29-38. doi: 10.7326/M22-1543. Epub 2022 Dec 20. PMID 36534976
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Davison SN. End-of-life care preferences and needs: perceptions of patients with chronic kidney disease. Clin J Am Soc Nephrol. 2010 Feb;5(2):195-204. doi: 10.2215/CJN.05960809. Epub 2010 Jan 14. PMID 20089488
- [Background] Reilly KL, Kennedy S, Porter G, Estabrooks P. Comparing, Contrasting, and Integrating Dissemination and Implementation Outcomes Included in the RE-AIM and Implementation Outcomes Frameworks. Front Public Health. 2020 Sep 2;8:430. doi: 10.3389/fpubh.2020.00430. eCollection 2020. PMID 32984239
- [Background] Wong SPY, McFarland LV, Liu CF, Laundry RJ, Hebert PL, O'Hare AM. Care Practices for Patients With Advanced Kidney Disease Who Forgo Maintenance Dialysis. JAMA Intern Med. 2019 Mar 1;179(3):305-313. doi: 10.1001/jamainternmed.2018.6197. PMID 30667475
- [Background] Morton RL, Tong A, Howard K, Snelling P, Webster AC. The views of patients and carers in treatment decision making for chronic kidney disease: systematic review and thematic synthesis of qualitative studies. BMJ. 2010 Jan 19;340:c112. doi: 10.1136/bmj.c112. PMID 20085970
- [Background] Murtagh FEM, Burns A, Moranne O, Morton RL, Naicker S. Supportive Care: Comprehensive Conservative Care in End-Stage Kidney Disease. Clin J Am Soc Nephrol. 2016 Oct 7;11(10):1909-1914. doi: 10.2215/CJN.04840516. Epub 2016 Aug 10. PMID 27510453
- [Background] Saeed F, Ladwig SA, Epstein RM, Monk RD, Duberstein PR. Dialysis Regret: Prevalence and Correlates. Clin J Am Soc Nephrol. 2020 Jul 1;15(7):957-963. doi: 10.2215/CJN.13781119. Epub 2020 Jun 4. PMID 32499230
- [Background] Chandna SM, Da Silva-Gane M, Marshall C, Warwicker P, Greenwood RN, Farrington K. Survival of elderly patients with stage 5 CKD: comparison of conservative management and renal replacement therapy. Nephrol Dial Transplant. 2011 May;26(5):1608-14. doi: 10.1093/ndt/gfq630. Epub 2010 Nov 22. PMID 21098012
- [Background] USRDS. USRDS Annual Data Report USRDS Annual Data Report. Chapter 1: Incidence, Prevalence, Patient Characteristics, and Treatment Modalities, United States Renal Data System. 2018. 42.
- [Background] Gale RC, Wu J, Erhardt T, Bounthavong M, Reardon CM, Damschroder LJ, Midboe AM. Comparison of rapid vs in-depth qualitative analytic methods from a process evaluation of academic detailing in the Veterans Health Administration. Implement Sci. 2019 Feb 1;14(1):11. doi: 10.1186/s13012-019-0853-y. PMID 30709368
- [Background] Rhodes T, Stimson GV, Fitch C, Ball A, Renton A. Rapid assessment, injecting drug use, and public health. Lancet. 1999 Jul 3;354(9172):65-8. doi: 10.1016/S0140-6736(98)07612-0. No abstract available. PMID 10406380
- [Background] Lupu DE, Aldous A, Anderson E, Schell JO, Groninger H, Sherman MJ, Aiello JR, Simmens SJ. Advance Care Planning Coaching in CKD Clinics: A Pragmatic Randomized Clinical Trial. Am J Kidney Dis. 2022 May;79(5):699-708.e1. doi: 10.1053/j.ajkd.2021.08.019. Epub 2021 Oct 12. PMID 34648897
- [Background] Teerenstra S, Eldridge S, Graff M, de Hoop E, Borm GF. A simple sample size formula for analysis of covariance in cluster randomized trials. Stat Med. 2012 Sep 10;31(20):2169-78. doi: 10.1002/sim.5352. Epub 2012 Apr 11. PMID 22495809
- [Background] Carson RC, Juszczak M, Davenport A, Burns A. Is maximum conservative management an equivalent treatment option to dialysis for elderly patients with significant comorbid disease? Clin J Am Soc Nephrol. 2009 Oct;4(10):1611-9. doi: 10.2215/CJN.00510109. Epub 2009 Sep 24. PMID 19808244
- [Background] Morton RL, Webster AC, McGeechan K, Howard K, Murtagh FEM, Gray NA, Kerr PG, Germain MJ, Snelling P. Conservative Management and End-of-Life Care in an Australian Cohort with ESRD. Clin J Am Soc Nephrol. 2016 Dec 7;11(12):2195-2203. doi: 10.2215/CJN.11861115. Epub 2016 Oct 3. PMID 27697783
- [Background] Saeed F, Schell JO. Shared Decision Making for Older Adults: Time to Move Beyond Dialysis as a Default. Ann Intern Med. 2023 Jan;176(1):129-130. doi: 10.7326/M22-3431. Epub 2022 Dec 20. No abstract available. PMID 36534979
- [Background] Korevaar E, Kasza J, Taljaard M, Hemming K, Haines T, Turner EL, Thompson JA, Hughes JP, Forbes AB. Intra-cluster correlations from the CLustered OUtcome Dataset bank to inform the design of longitudinal cluster trials. Clin Trials. 2021 Oct;18(5):529-540. doi: 10.1177/17407745211020852. Epub 2021 Jun 4. PMID 34088230
- [Background] Voldal EC, Hakhu NR, Xia F, Heagerty PJ, Hughes JP. swCRTdesign: An RPackage for Stepped Wedge Trial Design and Analysis. Comput Methods Programs Biomed. 2020 Nov;196:105514. doi: 10.1016/j.cmpb.2020.105514. Epub 2020 May 21. PMID 32554025
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Wongrakpanich S, Susantitaphong P, Isaranuwatchai S, Chenbhanich J, Eiam-Ong S, Jaber BL. Dialysis Therapy and Conservative Management of Advanced Chronic Kidney Disease in the Elderly: A Systematic Review. Nephron. 2017;137(3):178-189. doi: 10.1159/000477361. Epub 2017 May 25. PMID 28538218
- [Background] Buur LE, Madsen JK, Eidemak I, Krarup E, Lauridsen TG, Taasti LH, Finderup J. Does conservative kidney management offer a quantity or quality of life benefit compared to dialysis? A systematic review. BMC Nephrol. 2021 Sep 11;22(1):307. doi: 10.1186/s12882-021-02516-6. PMID 34507554
- [Background] Seow YY, Cheung YB, Qu LM, Yee AC. Trajectory of quality of life for poor prognosis stage 5D chronic kidney disease with and without dialysis. Am J Nephrol. 2013;37(3):231-8. doi: 10.1159/000347220. Epub 2013 Mar 2. PMID 23467046
- [Background] Foote C, Kotwal S, Gallagher M, Cass A, Brown M, Jardine M. Survival outcomes of supportive care versus dialysis therapies for elderly patients with end-stage kidney disease: A systematic review and meta-analysis. Nephrology (Carlton). 2016 Mar;21(3):241-53. doi: 10.1111/nep.12586. PMID 26265214
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Galla JH. Clinical practice guideline on shared decision-making in the appropriate initiation of and withdrawal from dialysis. The Renal Physicians Association and the American Society of Nephrology. J Am Soc Nephrol. 2000 Jul;11(7):1340-1342. doi: 10.1681/ASN.V1171340. No abstract available. PMID 10864592
- [Background] Koch-Weser S, Kennefick K, Tighiouart H, Wong JB, Gordon EJ, Isakova T, Rifkin D, Rossi A, Weiner DE, Ladin K. Development and Validation of the Rating of CKD Knowledge Among Older Adults (Know-CKD) With Kidney Failure. Am J Kidney Dis. 2024 May;83(5):569-577. doi: 10.1053/j.ajkd.2023.09.024. Epub 2023 Dec 7. PMID 38070590
- [Background] Wong SP, Kreuter W, O'Hare AM. Treatment intensity at the end of life in older adults receiving long-term dialysis. Arch Intern Med. 2012 Apr 23;172(8):661-3; discussion 663-4. doi: 10.1001/archinternmed.2012.268. No abstract available. PMID 22529233

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT06243068/Prot_SAP_ICF_002.pdf